CLINICAL TRIAL: NCT07253038
Title: The Social-HD Study: A Cross-Sectional Observational Study of Social Cognition in Early Huntington Disease
Brief Title: Evaluation of Three Tests to Assess Social Cognition in Huntington Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-04424-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Huntington Disease
Keywords: social cognition; apathy; cognition; depression; total functional capacity; total motor score
MeSH Terms: conditions — Huntington Disease; Lethargy; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Huntington disease: Participants with early Huntington disease
- Controls: Participants with no heritage of HD or negative pre-symptomatic HD gene test

SUMMARY:
The goal of this observational study is to learn about the usefulness of a test of social functioning in persons with Huntington disease. Huntington disease affects motor function, psychological well-being and cognitive functions ("thinking abilities" such as paying attention, remembering and solving problems). It is also believed to affect important social functions, including the ability to understand others' intentions and emotions (social cognition). The test of interest in this study is called The Double Movie for the Assessment of Social Cognition-Multiple Choice (DMASC-MC) and will be compared to two other similar and well-known tests. The main question which the study aims to answer is:

• Is DMASC-MC a useful tool for detecting problems with social functioning in adult persons with early Huntington disease? In the study, participants will meet with a medical doctor and a psychologist for assessment of different symptoms related to Huntington disease, including social functioning. Better methods for identifying problems with social functioning could help persons with Huntington disease and their families in mainly two ways. Firstly, it could increase their understanding of how the disease has affected them. Secondly, a better understanding of these problems could lead to better recommendations and interventions from medical teams, which would also benefit persons with Huntington disease and families.

DETAILED DESCRIPTION:
Background:

Huntington disease (HD) is a fatal neurodegenerative disorder that leads to motor disturbances, psychiatric symptoms and dementia. It is caused by an expanded CAG repeat in the huntingtin (HTT) gene which is inherited in an autosomal dominant fashion with full penetrance. It typically manifests in midlife. There are no disease-modifying therapies and current care is focused on reducing symptoms and improving quality of life. An important understudied part of the clinical manifestation is the early development of personality changes that have major impact on most aspects of the life of the affected person. These changes may be due to altered social cognition. Today, assessment of social cognition is often not part of the neuropsychological battery for HD and the so far investigated tests may not capture sufficient aspects of altered social cognition.

Aim:

The aim is to investigate whether the social cognitive test "Double Movie for the Assessment of Social Cognition-Multiple Choice (DMASC-MC) " will detect a significant difference in persons with early stages of HD compared to age and sex matched controls.

Methods:

This clinical research study will include 20 persons with early HD and 20 matched controls. The number of participants is based on a power calculation. The research participants will be assessed using DMASC-MC as well as two other tests for social cognition, Reading the Mind in the Eyes Test and The Emotion Hexagon Test. They will also be evaluated for typical cognitive deficits, psychiatric symptoms and motor aspects in HD.

Relevance:

This study aims to bridge an important gap in clinical care where evaluation of social cognition is not yet part of standard assessments. Determination of social cognitive deficits will be important for planning care and facilitate communication for HD families.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for persons with HD

1. Clinical diagnosis of HD
2. CAG repeat: 40 and more

Inclusion criteria for control group

1. No heritage of HD or negative pre-symptomatic HD gene test

Exclusion Criteria:

Participants in both groups are excluded from the study if any of the following criteria apply:

1. Dementia or MOCA<19, The Mini Mental State Examination (MMSE) <19
2. Other neurological disorders
3. Ongoing psychosis
4. Ongoing alcohol/drug addiction
5. Other native language than Swedish
6. Severe problems with vision and hearing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment of participants will be made at the HD clinic in Lund, Sweden and through ethical review board-approved advertisment material posted at social media platforms and websites hosted by the Huntingtoncenter at Lund and the Swedish patient organization Riksförbundet för Huntingtons sjukdom (RHS) as well as YTAN.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Significant difference in mean value of "Double Movie for the Assessment of Social Cognition-Multiple Choice" (DMASC-MC) total score between HD and controls | Baseline
  To investigate if persons with HD have a significantly lower score than a control group in the test "Double Movie for the Assessment of Social Cognition-Multiple Choice" (DMASC-MC)". DMASC-MC: Minimum value 0, maximum value 44, higher scores mean a better outcome.

SECONDARY OUTCOMES:
Significant difference in mean value of Reading the Mind in the Eyes Test (RMET) total score between HD and controls | Baseline
  To investigate if persons with HD have a significantly lower score than a control group in the Reading the Mind in the Eyes Test (RMET) test. RMET: Minimum value 0, maximum value 36, higher scores mean a better outcome.
Significant difference in mean value of Emotional Hexagon Test (EHT) total score between HD and controls | Baseline
  To evaluate if persons with HD have a significantly lower score than a control group in the Emotional Hexagon Test (EHT). EHT: Minimum value 0, maximum value 24, higher scores mean a better outcome.
Significant correlation between social cognitive test scores and Montreal Cognitive Assessment (MOCA) scores | Baseline
  To investigate if there is a correlation between social cognitive test scores and Montreal Cognitive Assessment (MOCA scores = cognitive scores). MOCA scale: Minimum value 0, maximum value 30 points, lower scores mean a worse outcome.
Significant correlation between social cognitive test scores and total functional capacity (TFC) scores | Baseline
  To investigate if there is a correlation between social cognitive test scores and total functional capacity (TFC scores =scores for everyday life function in HD). TFC: Minimum value 0, maximum value 13, higher scores mean a better outcome.
Significant correlation between social cognitive test scores and CAG-Age-Product (CAP) scores | Baseline
  To investigate if there is a correlation between social cognitive test scores and CAG-Age-Product (CAP scores =scores for disease burden).CAP scores are calculated as the product of the length of the expanded CAG repeat and age, indicating a cumulative burden that predicts progression of HD. Higher CAP product means larger disease burden.
Significant correlation between social cognitive test scores and total motor scores (TMS). | Baseline
  To investigate if there is a correlation between social cognitive test scores and total motor scores (TMS = motor scores). TMS: minimum value 0, maximum value 124, lower scores mean a better outcome.
Significant correlation between social cognitive test scores and Montgomery-Åsberg Depression Rating Scale (MADRS) scores | Baseline
  To investigate if there is a correlation between social cognitive test scores and Montgomery-Åsberg Depression Rating Scale (MADRS) scores (= depression scores). MADRS: Minimum value 0, maximum value 60, lower scores mean a better outcome.
Significant correlation between social cognitive test scores and apathy evaluation scale (AES) scores | Baseline
  To investigate if there is a correlation between social cognitive test scores and apathy evaluation scale (AES) scores (= apathy scores). AES: Minimum value 18, maximum value 72, lower scores mean a better outcome.
Significant correlation between social cognitive test scores and cognitive scores | Baseline
  To investigate if there is a correlation between social cognitive test scores and Symbol digit modalities test (SDMT)/D-KEFS Color Word Interference Test (CWIT)/ D-KEFS Verbal Fluency Test (VFT) scores (= cognitive scores). SDMT: Minimum value 0, maximum value 110, higher scores mean a better outcome.
  CWIT: no minimum value, maximum value 180, lower scores mean a better outcome. VFT: Minimum value 0, no maximum value, higher scores mean a better outcome.
Proportion of both HD subjects and control subjects with impaired results on each of the social cognitive tests, compared to norms. | Baseline
  Percentage of subjects within the HD group performing below 1,5 SD compared to norm data on DMASC-MC, RMET and EHT, compared to prior norm data. Percentage of subjects within the control group performing below 1,5 SD compared to norm data on DMASC-MC, RMET and EHT.

CONTACTS AND LOCATIONS:
Overall Officials: Asa Petersen, MD PhD, Principal Investigator — Department of Psychiatry, Skåne University Hospital
Locations (1):
- Skane University Hospital, Region Skane, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Home page for the Huntington Disease Center at Region Skate — https://huntingtoncentrum.se/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT07253038/Prot_SAP_000.pdf